CLINICAL TRIAL: NCT02225886
Title: Effects of Ascorbic Acid Administration in the Treatment of Anemia in Chronic Hemodialysed Patients With Iron Overload
Brief Title: Ascorbic Acid Administration in the Treatment of Anemia in Chronic Hemodialysed Patients
Acronym: FeVitC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anemia Working Group Romania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AWGRO 06/2014
Record Dates: First submitted 2014-08-23; First posted 2014-08-26 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Anaemia Response to the Treatment; Peripheral Iron Indices; Oxalemia
Keywords: Renal anaemia; Intravenous ascorbic acid; Intravenous iron administration
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ascorbic acid (Experimental): Patients will receive a 300 mg intravenous ascorbic acid, 3 times a week, postdialysis, except for the dialysis sessions when iv iron is administered.
  Interventions: Drug: Ascorbic Acid
- Control group (Placebo Comparator): Patients will receive 100 mL saline solution, 3 times a week, with associated medication, except but the dialysis sessions when iv iron is administered.
  Interventions: Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Ascorbic Acid — 300 mg of intravenous ascorbic acid will be given 3 times a week, postdialysis, in 100 mL saline solution, except for the dialysis sessions when iv iron is administered

SUMMARY:
The administration of ascorbic acid seemed to increase the iron available for erythropoiesis, thus improving the anemia response to the treatment.

The investigators therefore aimed to evaluate the effects of intravenous ascorbic acid administration in hemodialysed patients with iron overload.

DETAILED DESCRIPTION:
Renal anemia is a complex condition in which chronic inflammation, among other factors, can change the iron distribution by locking it in deposits, and also, iron metabolism parameters. Thus, is hard to separate the iron functional deficit from overload.

The ascorbic acid is a hydrosoluble vitamin capable of reduction and hydrolysis. As a reduction agent, the ascorbic acid supports the transformation of ferric iron to ferrous iron. For instance, the ascorbic acid can increase digestive absorption and taking over the iron without transferrin, helps iron release from ferritin and hemosiderin and delays ferritin conversion to hemosiderin; therefore, the administration of ascorbic acid can increase the quantity of iron available for erythropoiesis by realising it from the deposits.

Consequently, the antioxidant function of ascorbic acid can increase the red cells' lifetime, reducing the inflammation and improving erythropoietin response Following these premises, recent studies have examined the effect of administrating ascorbic acid to hemodialysed patients with erythropoiesis stimulating agents (ESA) hyporesponsiveness anemia and functional deficit or iron overload markers. The results of administering ascorbic acid revealed an increased level of hemoglobin and transferrin saturation (TSAT) combined with the decrease of ESA doses. The major limitations of these studies are the short amount of time for observation (<6months) and the limited number of participants which hampered neither the complete evaluation of the goals, nor the adverse effects of supplementary administration of vitamin C.

Until now, the Clinical practice guidelines of Kidney Disease do not recommend currently using of high doses of vitamin C, considering the risk of a high level of oxalemia and the limited information about the benefits. Considering this background, we intended to evaluate the benefits of intravenous administration of ascorbic acid in hemodialysed patients with iron balance markers suggestive for iron overload.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old
* At least 6 months on hemodialysis at the time of randomization;
* Kt/V≥1.2;
* average of the last three serum ferritin levels > 500 ng/mL AND
* Average of the last three TSAT levels > 20% and increasing
* ERI in the 4th quartile of the group

Exclusion Criteria:

* Active bleeding or other cause of anemia
* Serum level of intact parathyroid hormone (iPTH)>800 pg/mL
* Actual neoplasia
* HIV, Hepatitis B or C infections
* Significant inflammation (CRP>12mg/L) or acute infection
* Venous central catheter
* Severe hepatic, cardiovascular, psychic disease or other severe comorbidities
* Moderate or severe malnutrition
* Blood transfusions in the 2 months prior to screening
* Pregnancy or breastfeeding
* Inclusion in another clinical trial in the past month

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Variation of erythropoetin resistance index (ERI) | 12 months
  Erythropoietin resistance index: the dose of ESA divided by the level of Hb - will be calculated monthly.

SECONDARY OUTCOMES:
Percentage of patients with Hb in the target range | 12 months
  Percentage of patients with stable the hemoglobin in the target range (10.5-12g/dL), without any change in the weekly dose of ESA
Changes in ESA dose | 12 months
  The number of reductions or increases in the ESA dose during the study
Variation in ESA dose | 12 months
  The difference between the actual ESA dose and the one at baseline will be calculated monthly.
Variation of iron dose | 12 months
  The difference between the actual iron dose and the one at baseline will be calculated monthly.
Percentage of patients with hemoglobin within target | 12 months
  Percentage of patients with 10<Hb<12.1 g/dL will be calculated monthly.
Percentage of patients with target iron status | 12 months
  Percentage of patients with 100<serum ferritin<800 ng/mL and 19<transferrin saturation<51% will be calculated monthly.
Variation of serum hepcidin | 12 months
  Variation of serum hepcidin will be calculated every 3 months
Oxalemia | 12 months
  Serum oxalate level will be calculated every 3 months
Local and general tolerance to vitamin C | 12 months
  Local and general tolerance to vitamin C will be evaluated monthly
Adverse events | 12 months
  Adverse events will be evaluated monthly
The number of withdrawals and dropouts | 12 months
  The number of withdrawals and dropouts will be calculated monthly

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Mircescu, Professor, Study Chair — Anemia Working Group Romania; Liliana Garneata, MD, PhD, Study Director — Anemia Workiing Group Romania; Tudor Simionescu, MD, PhD, Principal Investigator — "Carol Davila" Teaching Hospital of Nephrology
Locations (1):
- "Nefrolab" Dialysis Center, Slatina, Romania

IPD SHARING:
Plan to Share IPD: Yes
Publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 24 months

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745